CLINICAL TRIAL: NCT01056094
Title: Effects of Lutein Supplementation on Oxidative Stress and Inflammation in Healthy Nonsmokers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Le MA, Xi'an Jiaotong University College of Medicine, Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNS-06094
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2009-04

CONDITIONS: Oxidative Stress in Healthy Subjects
MeSH Terms: interventions — Lutein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 20mg Lutein (Active Comparator): Dietary Supplement: 20mg Lutein; daily supplementation 12 week
  Interventions: Drug: Lutein
- 10mg Lutein (Active Comparator): Dietary Supplement: 10mg Lutein; daily supplementation 12 week
  Interventions: Drug: Lutein
- 0mg Lutein (Placebo Comparator): Dietary Supplement: 0mg Lutein; daily supplementation 12 week
  Interventions: Drug: Lutein

INTERVENTIONS:
Drug: Lutein — Dietary Supplement: 20mg,10mg, 0mg Lutein; daily supplementation 12 week

SUMMARY:
Lutein is one of oxygenated carotenoids. Over the past few years, there has been increased interest in evaluating the effect of lutein for optimizing immune functions. A large number of epidemiological studies support the notion that a high intake of lutein is associated with a reduced risk of coronary heart disease and certain types of cancer. The biological mechanisms for the protective effects of this carotenoid, including powerful modulation of functions and antioxidant properties, are only partially known. Although several nutrients and phytochemicals have been shown to modulate immune functions in humans, few studies have investigated the role of lutein consumption. No information is available as to whether lutein supplementation could be protective against oxidative stress. Therefore, the objective of the present study was to examine the effect of consuming different doses of lutein on oxidative stress in healthy subjects.

DETAILED DESCRIPTION:
Participants with a history of smoking, alcohol consumption, body mass index (BMI)≥30kg/m2, allergies, ocular diseases and participants taking vitamins or other food supplements containing lutein were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects aged in the range of 20 to 80

Exclusion Criteria:

* Participants with a history of smoking
* Alcohol consumption
* Body mass index (BMI)≥30kg/m2
* Allergies
* Ocular diseases or recent infections(within the last year) and participants taking vitamins or other food supplements containing lutein the previous 2 months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-07 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of lipid, protein and DNA oxidative damage, marker of antioxidant capacity and antioxidant enzyme activities(GPx,SOD and CAT)in healthy subjects. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Xi'an Jiaotong University College of Medicine, Xi'an, Shaanxi, China